CLINICAL TRIAL: NCT04124848
Title: Evaluating the Prevalence and Implications of Obstructive Sleep Apnea Among Somali-Americans: A Translational Research Study
Brief Title: Obstructive Sleep Apnea Among Somali-Americans
Acronym: Somali OSA
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Sleep Number Corporation (Unknown)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: 19-000033
Record Dates: First submitted 2019-10-07; First posted 2019-10-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Somali-Americans; Sleep Disordered Breathing; Cardiovascular Diseases; Sex and Racial Differences; Respiratory Disorders; Hypertension; Diabetes; Health Disparities
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Cardiovascular Diseases; Coitus; Respiration Disorders; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma, buffy coat, and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Somali Descent: Study participants who are of Somali origin.
- Non-Somali Descent: Study participants who are not of Somali origin.

SUMMARY:
The investigators seek to advance the understanding of obstructive sleep apnea as it relates to different ethnic origins as well as sex differences. The investigators will compare Somali patients with known obstructive sleep apnea (OSA) to individuals without OSA, and to individuals of other ethnic/racial origins to determine the risk factors (genetic and/or physiologic) associated with developing cardiovascular diseases. This will help the investigators to understand the unique sleep pathology of individuals of African descent.

DETAILED DESCRIPTION:
Participants can be healthy volunteers or volunteers diagnosed with obstructive sleep apnea. All patients may undergo a sleep study (i.e. hospital or home-based), physical examination, questionnaires, blood and urine samples, ultrasound scan of the heart and brachial artery in the arm, CT scan, DEXA scan, paced breathing test, cardiopulmonary test and chemo-sensitivity test.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Somali, African, Asian, and European descent.
* Adult males and females who are older than 18 years of age.

Exclusion Criteria:

* Minors under 18 years or adults over 100 years
* Positive pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are individuals who are of Somali descent compared to those of different racial/ethnic origins.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of obstructive sleep apnea | 10 years
  Measure the apnea-hypopnea index (AHI) to determine burden of obstructive sleep apnea. Based on the AHI, sleep apnea will be diagnosed if the AHI is ≥5 events/hour.
To determine the severity of obstructive sleep apnea | 10 years
  The severity of OSA is classified based on the AHI as follows: None/Minimal: AHI < 5 per hour, Mild: AHI ≥ 5, but < 15 per hour, Moderate: AHI ≥ 15, but < 30 per hour, Severe: AHI ≥ 30 per hour.

SECONDARY OUTCOMES:
24 hour mean arterial pressure | 10 years
  Ambulatory measure of blood pressure in mmHg
Vascular endothelial function | 10 years
  Change in brachial artery diameter in response to hyperemia
Insulin sensitivity | 10 years
  Oral glucose tolerance testing
Body composition | 10 years
  Percentage body fat content

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenlund IM, Bock JM, Govindan N, Kantas D, Singh P, Covassin N, Somers VK. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. J Racial Ethn Health Disparities. 2025 Mar 15:10.1007/s40615-025-02389-7. doi: 10.1007/s40615-025-02389-7. Online ahead of print. PMID 40088388
- [Derived] Greenlund I, Bock J, Govindan N, Kantas D, Singh P, Covassin N, Somers V. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. Res Sq [Preprint]. 2024 Oct 21:rs.3.rs-4925722. doi: 10.21203/rs.3.rs-4925722/v1. PMID 39502777